CLINICAL TRIAL: NCT05925218
Title: Circulating Tumor DNA Collection From Patients With High Grade Gliomas
Acronym: m-ctDNA
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5047
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy as per standard of care — Adjuvant Radiotherapy +/- systemic therapy as per standard of care

SUMMARY:
Improved outcomes for high-grade gliomas (HGG) require advances in our ability to monitor changes to tumour biology using non-surgical approaches. "Liquid biopsy" is a term used to describe a technique whereby tumour DNA, which has been shed off and then circulates through the blood stream, is detected and analyzed. Our goal is to develop a new type of liquid biopsy that is suitable for primary brain tumours that uses a method that is highly sensitive and allows for ongoing analysis of these tumours.

DETAILED DESCRIPTION:
The study objective is to determine the feasibility of measuring both the burden and key molecular features of HGG through profiling of plasma circulating tumour DNA (ctDNA). This will be determined by detecting ctDNA in samples from HGG patients, and measuring changes in ctDNA levels over time following HGG treatment. 50 eligible patients will be enrolled in the study at University Health Network, and up to 10 blood samples will be obtained; up to 2 blood samples prior to their radiotherapy treatment, and 8 blood samples after their radiotherapy treatment. If available, tissue samples that are stored at UHN will also be collected for DNA extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients can be enrolled either prior to a planned surgery/biopsy for a suspected HGG or after biopsy/surgery of pathologically proven, previously untreated HGG, prior to adjuvant radiotherapy
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Age ≥18 yrs

Exclusion Criteria:

* History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for ≥ 2 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or pathologically-proven, previously untreated high grade gliomas
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of measuring both the burden and key molecular features of high- grade gliomas (HGG) through profiling of plasma circulating tumour DNA (ctDNA) | 2 years
  Feasibility in this context will be defined by 1) detecting ctDNA in samples from HGG patients and 2) measuring changes in levels of specific ctDNA fragments following HGG treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share.